CLINICAL TRIAL: NCT02726373
Title: The Effect of Intermittent vs. Continuous Walking Training on Walking Endurance and Fatigue in People With Multiple Sclerosis: a Randomized, Crossover Trial.
Brief Title: Comparison of Intermittent vs. Continuous Walking in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Herb Karpatkin, Assistant Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INTCON1
Record Dates: First submitted 2016-03-30; First posted 2016-04-01 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Sclerosis, Endurance
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent walking training (Experimental)
  Interventions: Other: type of walking
- Continuous Walking Training (Active Comparator)
  Interventions: Other: type of walking

INTERVENTIONS:
Other: type of walking — Subjects walked either intermittently or continuously twice a week for 4 weeks, then crossed over

SUMMARY:
Objective: To compare effects of an intermittent and continuous walking program on walking endurance and fatigue in people with multiple sclerosis (MS).A randomized crossover prospective method was used.The intervention consisted of eight 6-minute-long walks (2x/week for 4 weeks). The continuous condition consisted of 6 continuous minutes of walking. The intermittent condition consisted of three 2-minute bouts with 2-minute rests. After a 4-week detraining period, participants performed the second training condition.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnosis of MS
* Ambulatory for at least 6 minutes with or without an assistive device (e.g. cane, crutches or orthotics)
* Ability to read, understand, and sign an informed consent form

Exclusion Criteria:

* Evidence of exacerbation in the prior three months as defined by a treating physician
* Orthopedic or cardiovascular condition that would interfere with ability to walk for 6 continuous minutes,
* Currently being on an active physical rehabilitation program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pre to post change in 6 Minute walk test distance | 4 weeks

SECONDARY OUTCOMES:
Visual Analog Scale of fatigue | 4 weeks
  Measurements to be taken at baseline and after each 4 week intervention

IPD SHARING:
Plan to Share IPD: No